CLINICAL TRIAL: NCT02158364
Title: Freeze-dried Live Attenuated Measles and Rubella Combined Vaccine "Takeda" Specified Drug-use Survey of Vaccinees After the Second Vaccination
Brief Title: Freeze-dried Live Attenuated Measles/Rubella Combined Vaccine (Schwarz FF-8 Strain/TO-336 Strain) Specified Drug-use Survey of Vaccinees After the Second Vaccination
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 247-012; JapicCTI- 142507 (Registry Identifier: JapicCTI); JapicCTI-R171016 (Other: JapicCTI)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Measles/Rubella
Keywords: Pharmacological therapy
MeSH Terms: conditions — Measles; Rubella

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Live attenuated measles/rubella combined vaccine: Live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) is dissolved in 0.7 mL of accompanying reconstitution fluid (water for injection [Japanese Pharmacopoeia]), and a 0.5-mL portion is typically administered subcutaneously as a single dose.
  Interventions: Drug: Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain)

INTERVENTIONS:
Drug: Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) — Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain)
  Other Names: Freeze-dried live attenuated measles and rubella combined vaccine "Takeda"

SUMMARY:
The purpose of this survey is to assess the safety of freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) (freeze-dried live attenuated measles and rubella combined vaccine "Takeda") in terms of the occurrence of unknown/known adverse drug reactions and factors that may influence the safety of vaccinees after the second vaccination.

DETAILED DESCRIPTION:
This survey was designed to assess the safety of freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336strain) (freeze-dried live attenuated measles and rubella combined vaccine "Takeda") in terms of the occurrence of unknown/known adverse drug reactions and factors that may influence safety after the second vaccination.

Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) is dissolved in 0.7 mL of accompanying reconstitution fluid (water for injection [Japanese Pharmacopoeia]), wherein a 0.5-mL portion is typically administered subcutaneously as a single dose.

In addition, freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) should be used in accordance with the "Regulations for Vaccination" and the "Guidelines for Routine Vaccination."

ELIGIBILITY:
Inclusion Criteria:

-

Vaccinees who meet both of the following conditions [1] and [2]:

1. Vaccinees who have a prior history of receiving measles and/or rubella vaccination and who received freeze-dried live attenuated measles and rubella combined vaccine "Takeda" as the second vaccination
2. Vaccinees whose guardians are able to participate in a questionnaire survey on the health status of vaccinees after vaccination with freeze-dried live attenuated measles and rubella combined vaccine "Takeda"

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Measles/rubella
Sampling Method: Non-Probability Sample
Enrollment: 3331 (Actual)
Dates: Start 2007-03-28 (Actual); Primary Completion 2011-02-20 (Actual); Study Completion 2011-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 147 investigative sites in Japan, from 28-Mar-2007 to 20-Feb-2011.
Pre-assignment Details: Participants with a history of initial vaccination with live attenuated measles/rubella combined vaccine who received second vaccination with live attenuated measles/rubella combined vaccine as per routine medical practice were observed in this study.
Groups:
- Live Attenuated Measles/Rubella Combined Vaccine: Live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) is dissolved in 0.7 mL of accompanying reconstitution fluid (water for injection [Japanese Pharmacopoeia]), and a 0.5-mL portion is typically administered subcutaneously as a single dose. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Started | 3331
Completed | 3271
Not Completed | 60
Not completed — Case report forms uncollected | 10
Not completed — Protocol Deviation | 50

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All the enrolled participants who were completed the study without any protocol deviations and collected case report forms.
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3271
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1601
  Male | 1670
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 3271
Predisposition to Hypersensitivity [Count of Participants; unit: Participants]
  Had Predisposition to Hypersensitivity | 403
  Had no Predisposition to Hypersensitivity | 2868
Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Complications | 257
    Had No Complications | 3014
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had Medical History | 492
    Had No Medical History | 2779
Concurrent Medication [Count of Participants; unit: Participants]
  Had Concurrent Medication(s) | 169
  Had No Concurrent Medication | 3099
  Unknown/not reported | 3
Cautions to Vaccination [Count of Participants; unit: Participants]
  Had Cautions | 169
  Had no Cautions | 3102
History of Vaccination with Measles Vaccine [Count of Participants; unit: Participants]
  Received the Vaccine | 2902
  Unknown/not reported | 369
History of Vaccination with Rubella Vaccine [Count of Participants; unit: Participants]
  Received the Vaccine | 2871
  Unknown/not reported | 400
History of Vaccination with Measles/Rubella Combined Vaccine [Count of Participants; unit: Participants]
  Received the Vaccine | 351
  Unknown/not reported | 2920
Type of Surveying Method after Vaccination [Number; unit: Participants] — Type of surveying method after vaccination included questionnaire, consultation and other survey (for example, call). Participants may be represented in more than 1 category.
  Participants
    Questionnaire, Available | 3023
    Questionnaire, not Available | 248
    Physician's Visit, Yes | 653
    Physician's Visit, No | 2618
    Other, Yes | 147
    Other, No | 3124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Drug Reactions (ADRs)
Description: Serious ADRs are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Frequency of adverse events and factors that may influence safety were not to be assessed as endpoints of this study and were registered as endpoints by mistake. Instead, ADRs were assessed as endpoint.
Time Frame: Up to Day 28
Population: Vaccinated Safety Analysis Set included all participants who received measles/rubella combined vaccine "Takeda" as the second vaccination. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3225
Participants | 2

2. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AE are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3225
Participants | 590

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Serious Adverse Events (participants affected / at risk) | 2/3225
Other Adverse Events (participants affected / at risk) | 376/3225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Live Attenuated Measles/Rubella Combined Vaccine (N=3225)
Convulsion (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Live Attenuated Measles/Rubella Combined Vaccine (N=3225)
Injection site erythema (General disorders) | 214
Pyrexia (General disorders) | 162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.